CLINICAL TRIAL: NCT02476266
Title: Power Training to Reduce Falls in Parkinson's Disease
Brief Title: Two Resistance Training Protocols to Reduce the Risk of Falls in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Life Financial Movement Disorders Research and Rehabilitation Centre (Other)
Responsible Party: Principal Investigator, Brittany Intzandt, Graduate Student, Sun Life Financial Movement Disorders Research and Rehabilitation Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3992
Record Dates: First submitted 2015-06-16; First posted 2015-06-19 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Parkinson's Disease; Accidental Falls
Keywords: resistance training; strength training; balance; muscle strength
MeSH Terms: conditions — Parkinson Disease | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Participants randomized to this group will come in for testing at pre-intervention, post-intervention, three month wash out and six month wash out. Participants will be asked to continue their activities of daily living. To account for any physical activity changes over the length of the study the Community Healthy Activities Model Program for Seniors (CHAMPS) questionnaire will be administered to all individuals. A control group is necessary to compare to show normal disease progression over the length of the study as well as to demonstrate that improvements in outcome measures are due to the interventions and not practice effects.
- Strength Training (Active Comparator): Individuals randomized to this program will complete three sets of eight to ten repetitions at 70% of their predicted 1-RM for each of the exercises mentioned above. The speed of the movements in this program will be two to three seconds each for the concentric and eccentric components. When participants are able to complete ten repetitions in their third set for two consecutive days, weight will be increased for the following session by 5% of the current weight that they are at in accordance with Canadian Society for Exercise Physiology (CSEP) and American College of Sports Medicine (ACSM) guidelines. Participants will complete a total of 24 sessions over the course of 12 weeks, two times per week for an hour each session.
  Interventions: Other: Resistance Training
- Power Training (Experimental): Participants randomized to this program will complete three sets of 12 to 15 repetitions completed at 40% of predicted 1-RM for each exercises. The concentric part of the movement will be completed as fast as possible, whereas the eccentric component will be accomplished in two to three seconds. The load in this group is lower as it has been shown that by performing power training at lighter loads, the muscles are able to be activated, throughout the entire concentric component, while maintaining a consistent level of force. The progression will be determined through the same means as the conventional strength training group. Participants will complete a total of 24 sessions over 12 weeks, twice per week for an hour each session
  Interventions: Other: Resistance Training

INTERVENTIONS:
Other: Resistance Training — Resistance training has been shown to improve balance and muscle weakness in those with PD as well as reducing the number of falls experienced, albeit not significantly. However to date no study has investigated forms of resistance training in the same study. To disentangle which form of resistance training might be more effective at reducing the risk of falls, improving balance and muscle strength, the proposed study will compare power training and conventional strength training.
  Arms: Power Training; Strength Training

SUMMARY:
Parkinson's disease (PD) is a chronic neurodegenerative disorder that is characterized by a multitude of symptoms. Impairments in balance, muscle deficits and increased risk of falls are commonly experienced in PD.The purpose of this study is to investigate the effects of two different resistance training programs on improving balance and muscular strength to thereby reduce the risk of falls in those with PD. This study will randomize individuals to one of two groups, a power training group, or a strength training group. Both interventional groups will participate in 12 weeks of resistance training, two times per week for an hour each exercise session.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder that results in multiple hallmark symptoms, such as balance impairments, postural instability and muscular deficits. These symptoms, in combination with a deficient sensory-perceptual integration system, put individuals with PD at a higher risk of falls and fractures, compared to healthy older adults. With the expected rise in PD diagnosis, this will place an unprecedented burden on the Canadian healthcare system due to increased hospitalizations, surgeries, placement into long term care facilities, and rehabilitation. Improving symptom severity and delaying disease progression through rehabilitation strategies that improve balance and muscular deficits, can decrease falling risk in individuals with PD, potentially alleviating the projected burden on the healthcare system. For these reasons it is imperative to have the ability to directly measure the degree to which individuals with PD are at risk of experiencing falls through objective techniques.

Purpose: Therefore the purpose of this study is to examine the effects of two different forms of resistance training (RT) to improve the muscular deficits experienced, as well to improve the balance impairments experienced as it has been suggested that RT is able to do this not only in healthy older adults but in those with PD as well. The two RT programs that will be investigated are a conventional strength training (ST) program and a high velocity strength training, known as power training (PT) program.

Objective/Aim: The objective of this study is to identify if ST or PT is a more effective rehabilitation program to improving muscle strength and power, balance measures and reducing the risk of falls. Due to the nature of the PT intervention it is hypothesized that these individuals will experience the greatest improvements in outcome measures.

Methods/Design: This study will be a double blind randomized controlled trial. Participants will be blinded to group allocation except for the control group, however those in the interventional group will only be informed that they are participating in a RT program. The primary investigator will only collect measures that are considered to be objective at follow up time points. Pre-intervention measures will all be collected prior to randomization into group allocations. The assessor of disease severity will also be blinded to group allocation.

Participants will be randomized to one of three groups: i) a control group (to account for normal disease progression for the duration of the intervention); ii) ST group and iii) PT group.

The intervention will be a total of 12 weeks long, where participants will come in two days per week for an hour long session each day, for a total of 24 session.

Participants randomized to the ST group will complete three sets of 8-10 repetitions at 70% of their one repetition maximum (1-RM), as determined during their pre-test. Those randomized to the PT group will complete three sets of 12-15 repetitions at 40% of their 1-RM, as determined during their pre-test. Both programs involve individualized exercise prescriptions based on the results of their predicted 1-RM. This program will be designed by a Canadian Society for Exercise Physiology Certified Exercise Physiologist, who has the knowledge and ability to safely test and prescribe exercise to individuals with chronic conditions. Both programs will be progressive in nature, in that as each individual is able to complete the last set, for two consecutive training sessions at the higher end of the range of repetitions (i.e. for the ST group 10 or more repetitions), the next session their weight will be increased by 5%. Upon completion participants will complete all outcome measures again. These measures will be completed during a wash out period at 3 months and 6 months post intervention to investigate the potential long term effects of these rehabilitation programs, and if either is more advantageous in the long term.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic PD by a Neurologist
* Able to stand two minutes, unassisted
* Able to understand English instructions
* Signed Physical Activity Readiness Medical Examination (PARmed-X) by physician

Exclusion Criteria:

* a neurological disease other than PD
* peripheral neuropathy
* physical impairments that would prevent participation in the muscular strength testing
* uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Lean-and-Release Perturbation Technique. | Change in muscle activity, compensatory postural responses from baseline to 12 weeks.
  This measure will require participants to be in a forward static lean at a maximum lean angle of 20 degrees from the vertical. This measure will induce a fall like situation where participants will be required to respond to this "perturbation" as they would in a slip or a trip scenario in real life. Muscle activity will be collected through surface electromyography (sEMG) to measure muscular responses associated with the perturbation. Measurement of postural adjustments will be made on an electronic carpet. sEMG and postural adjustments will demonstrate participants' onset of muscular activation time, latency to stepping, movement speed, and stepping characteristics.
Lean-and-Release Perturbation Technique. | Change in muscle activity, compensatory postural responses from 12 weeks to three month wash out
Lean-and-Release Perturbation Technique. | Change in muscle activity, compensatory postural responses from 12 weeks to six month wash out

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale Motor Subsection (UPDRS III) | Change in motor severity from baseline to 12 weeks
  Motor symptom severity as assessed by a movement disorders specialist
Unified Parkinson's Disease Rating Scale Motor Subsection (UPDRS III) | Change in motor severity from 12 weeks to three month wash out
Unified Parkinson's Disease Rating Scale Motor Subsection (UPDRS III) | Change in motor severity from 12 weeks to six month wash out
Gait Measurement | Changes in gait measures from baseline to 12 weeks
  This measures spatiotemporal gait parameters of individuals. This will allow measurement of key predictors of fall risk in PD, including step length, step time, step width, velocity, double support time, double support time percentage, step time variability, and step length variability. Participants will also perform a secondary digit-monitoring task while walking in the same well-lit open room. Participants will walk while simultaneously listening to an audio track of random numbers greater than zero and less than 10. For each trial that included this task, the participants are assigned two specific digits and will be instructed to silently count (without the use of manual aid) the number of times those two digits were announced by the audio track, separately. At the end of the trial the participants will be asked to inform the tester of the number of times they heard each digit.
Gait Measurement | Changes in gait measures from 12 weeks to three month wash out
  This measures spatiotemporal gait parameters of individuals. This will allow measurement of key predictors of fall risk in PD, including step length, step time, step width, velocity, double support time, double support time percentage, step time variability, and step length variability. Participants will also perform a secondary digit-monitoring task while walking in the same well-lit open room. Participants will walk while simultaneously listening to an audio track of random numbers greater than zero and less than 10. For each trial that included this task, the participants are assigned two specific digits and will be instructed to silently count (without the use of manual aid) the number of times those two digits were announced by the audio track, separately. At the end of the trial the participants will be asked to inform the tester of the number of times they heard each digit.
Gait Measurement | Changes in gait measures from 12 weeks to six month wash out
  This measures spatiotemporal gait parameters of individuals. This will allow measurement of key predictors of fall risk in PD, including step length, step time, step width, velocity, double support time, double support time percentage, step time variability, and step length variability. Participants will also perform a secondary digit-monitoring task while walking in the same well-lit open room. Participants will walk while simultaneously listening to an audio track of random numbers greater than zero and less than 10. For each trial that included this task, the participants are assigned two specific digits and will be instructed to silently count (without the use of manual aid) the number of times those two digits were announced by the audio track, separately. At the end of the trial the participants will be asked to inform the tester of the number of times they heard each digit.
Balance Measurement | Changes in postural stability measures from baseline to 12 weeks
  The Biodex Balance System™ SD will be used to assess balance outcomes. Specifically participants will be asked to complete two static balance tasks: i) eyes open- participants will be required to stand quietly for thirty seconds looking straight ahead and ii) eyes closed- participants will be required to stand quietly for thirty seconds with their eyes closed. Centre of pressure excursion will be measured in the anterior-posterior and medial-lateral directions to give an indication of participants overall postural stability.
Balance Measurement | Changes in postural stability measures from 12 weeks to three month wash out
  The Biodex Balance System™ SD will be used to assess balance outcomes. Specifically participants will be asked to complete two static balance tasks: i) eyes open- participants will be required to stand quietly for thirty seconds looking straight ahead and ii) eyes closed- participants will be required to stand quietly for thirty seconds with their eyes closed. Centre of pressure excursion will be measured in the anterior-posterior and medial-lateral directions to give an indication of participants overall postural stability.
Balance Measurement | Changes in postural stability measures from 12 weeks to six month wash out
  The Biodex Balance System™ SD will be used to assess balance outcomes. Specifically participants will be asked to complete two static balance tasks: i) eyes open- participants will be required to stand quietly for thirty seconds looking straight ahead and ii) eyes closed- participants will be required to stand quietly for thirty seconds with their eyes closed. Centre of pressure excursion will be measured in the anterior-posterior and medial-lateral directions to give an indication of participants overall postural stability.
Muscular Strength and Power Assessment | Changes in muscle strength measures from baseline to 12 weeks
  Technogym Selection Leg Press used to assess muscular strength and power. Participants will be completing a submaximal muscular strength protocol (multiple repetition maximum), which can be used to predict a one repetition maximum (1-RM).
Muscular Strength and Power Assessment | Changes in muscle strength measures from 12 weeks to three month wash out
  Technogym Selection Leg Press used to assess muscular strength and power. Participants will be completing a submaximal muscular strength protocol (multiple repetition maximum), which can be used to predict a one repetition maximum (1-RM).
Muscular Strength and Power Assessment | Changes in muscle strength measures from 12 weeks to six month wash out
  Technogym Selection Leg Press used to assess muscular strength and power. Participants will be completing a submaximal muscular strength protocol (multiple repetition maximum), which can be used to predict a one repetition maximum (1-RM).
Timed Up and Go (TUG) | Changes in time and gait measures from baseline to 12 weeks
  A timed up and go test (TUG test) will be administered as an assessment of function. Briefly, participants will be asked to begin the test by sitting in a chair, then to get up out of the chair without use of their hands and walk three metres then turn around and walk back to the chair and sit in it. Gait characteristics will be measured (step time, step length, step variability, velocity, time spent in double support. This test will occur three times.
Timed Up and Go (TUG) | Changes in time and gait measures from 12 weeks to three month wash out
  A timed up and go test (TUG test) will be administered as an assessment of function. Briefly, participants will be asked to begin the test by sitting in a chair, then to get up out of the chair without use of their hands and walk three metres then turn around and walk back to the chair and sit in it. Gait characteristics will be measured (step time, step length, step variability, velocity, time spent in double support. This test will occur three times.
Timed Up and Go (TUG) | Changes in time and gait measures from 12 weeks to six month wash out
  A timed up and go test (TUG test) will be administered as an assessment of function. Briefly, participants will be asked to begin the test by sitting in a chair, then to get up out of the chair without use of their hands and walk three metres then turn around and walk back to the chair and sit in it. Gait characteristics will be measured (step time, step length, step variability, velocity, time spent in double support. This test will occur three times.
Thirty Second Sit to Stand | Change in number of sit to stands completed from baseline to 12 weeks
  A thirty second sit to stand test will also be used as it is a functional measure of lower limb muscle strength. Participants will begin the test by sitting in a chair that is placed against a wall for safety. They will then be asked to go from a sitting position to a standing position as many times as possible in a thirty second time frame.
Thirty Second Sit to Stand | Change in number of sit to stands completed from 12 weeks to three month wash out
  A thirty second sit to stand test will also be used as it is a functional measure of lower limb muscle strength. Participants will begin the test by sitting in a chair that is placed against a wall for safety. They will then be asked to go from a sitting position to a standing position as many times as possible in a thirty second time frame.
Thirty Second Sit to Stand | Change in number of sit to stands completed from 12 weeks to six month wash out
  A thirty second sit to stand test will also be used as it is a functional measure of lower limb muscle strength. Participants will begin the test by sitting in a chair that is placed against a wall for safety. They will then be asked to go from a sitting position to a standing position as many times as possible in a thirty second time frame.

OTHER OUTCOMES:
Parkinson's disease Quality of Life Questionnaire (PDQ-39) | Change in score from baseline to 12 weeks
  It is one of the most widely used questionnaires to assess the quality of life of individuals with Parkinson's disease. For the purposes of this study it is imperative to identify if those that are at a higher risk of falling have a lower quality of life rating, as has been reported in previous studies. It is important to observe if the proposed measure that is to be validated is correlated with quality of life ratings.
CHAMPS Questionnaire | Changes in score from baseline to 12 weeks
  This questionnaire is able to quantify the amount of physical activity that older adults complete. This questionnaire is being used to control for varying activity levels, as it is proposed that those that have lower levels of physical activity are at a greater risk of falls. It is a self-administered questionnaire that takes approximately 10 to 15 minutes to complete. As well this questionnaire is important to administer, as participants will be asked to come in over a period of time, it is necessary to control and account for changes in physical activity levels that might influence the other outcome measures in this study.
CHAMPS Questionnaire | Changes in score from 12 weeks three month wash out
  This questionnaire is able to quantify the amount of physical activity that older adults complete. This questionnaire is being used to control for varying activity levels, as it is proposed that those that have lower levels of physical activity are at a greater risk of falls. It is a self-administered questionnaire that takes approximately 10 to 15 minutes to complete. As well this questionnaire is important to administer, as participants will be asked to come in over a period of time, it is necessary to control and account for changes in physical activity levels that might influence the other outcome measures in this study.
CHAMPS Questionnaire | Changes in score from 12 weeks six month wash out
  This questionnaire is able to quantify the amount of physical activity that older adults complete. This questionnaire is being used to control for varying activity levels, as it is proposed that those that have lower levels of physical activity are at a greater risk of falls. It is a self-administered questionnaire that takes approximately 10 to 15 minutes to complete. As well this questionnaire is important to administer, as participants will be asked to come in over a period of time, it is necessary to control and account for changes in physical activity levels that might influence the other outcome measures in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Intzandt, BSc, Study Director — Wilfrid Laurier University
Locations (1):
- Sunlife Financial Movement Disorders Research and Rehabilitation Centre- Wilfrid Laurier University, Waterloo, Ontario, Canada

REFERENCES:
- [Background] Glendinning DS, Enoka RM. Motor unit behavior in Parkinson's disease. Phys Ther. 1994 Jan;74(1):61-70. doi: 10.1093/ptj/74.1.61. PMID 8265729
- [Background] Stolze H, Klebe S, Baecker C, Zechlin C, Friege L, Pohle S, Deuschl G. Prevalence of gait disorders in hospitalized neurological patients. Mov Disord. 2005 Jan;20(1):89-94. doi: 10.1002/mds.20266. PMID 15390043
- [Background] Wielinski CL, Erickson-Davis C, Wichmann R, Walde-Douglas M, Parashos SA. Falls and injuries resulting from falls among patients with Parkinson's disease and other parkinsonian syndromes. Mov Disord. 2005 Apr;20(4):410-415. doi: 10.1002/mds.20347. PMID 15580552
- [Background] Newton RU, Murphy AJ, Humphries BJ, Wilson GJ, Kraemer WJ, Hakkinen K. Influence of load and stretch shortening cycle on the kinematics, kinetics and muscle activation that occurs during explosive upper-body movements. Eur J Appl Physiol Occup Physiol. 1997;75(4):333-42. doi: 10.1007/s004210050169. PMID 9134365
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886